CLINICAL TRIAL: NCT01428765
Title: GLORIA-AF: Global Registry on Long-Term Oral Anti-thrombotic TReatment In PAtients With Atrial Fibrillation (Phase I)
Brief Title: GLORIA-AF Registry Program (Phase I)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.114
Record Dates: First submitted 2011-08-25; First posted 2011-09-05 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
This study constitutes Phase I of the Registry Program. The main objective of this study is to characterize the newly diagnosed non-valvular AF patient population at risk for stroke and the selection of antithrombotic treatment for stroke prevention in a real-world setting before dabigatran etexilate is approved for the prevention of strokes and systemic emboli in patients with non-valvular AF in different regions of the world.

DETAILED DESCRIPTION:
Study Design:

cross-sectional

ELIGIBILITY:
Inclusion criteria:

1) Patients newly diagnosed with non-valvular atrial fibrillation at risk for stroke.

Exclusion criteria:

1. Presence of any mechanical heart valve, or valve disease that is expected to require valve replacement intervention;
2. Patients who have received more than 60 days of oral anticoagulant treatment (vitamin K antagonist) (VKA) in their lifetime;
3. Atrial fibrillation (AF) with a generally reversible cause;
4. Patients with a medical condition other than atrial fibrillation for which chronic use of an oral anticoagulant (VKAs) is indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with non-valvular atrial fibrillation at risk for stroke
Sampling Method: Non-Probability Sample
Enrollment: 1096 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (62):
- China (25):
  - 1160.114.08017 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.114.08018 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.114.08019 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.114.08020 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.114.08023 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.114.08024 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.114.08025 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.114.08007 Boehringer Ingelheim Investigational Site, Changsha
  - 1160.114.08021 Boehringer Ingelheim Investigational Site, Dalian
  - 1160.114.08004 Boehringer Ingelheim Investigational Site, Ghuangzhou
  - 1160.114.08006 Boehringer Ingelheim Investigational Site, Ghuangzhou
  - 1160.114.08001 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1160.114.08002 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1160.114.08005 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1160.114.08011 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1160.114.08015 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1160.114.08026 Boehringer Ingelheim Investigational Site, Nanjing
  - 1160.114.08010 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.114.08012 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.114.08014 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.114.08016 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.114.08027 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.114.08028 Boehringer Ingelheim Investigational Site, Shenzhen
  - 1160.114.08022 Boehringer Ingelheim Investigational Site, Tianjin
  - 1160.114.08008 Boehringer Ingelheim Investigational Site, Wuhan
- Croatia (4):
  - 1160.114.04002 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1160.114.04001 Boehringer Ingelheim Investigational Site, Opatija
  - 1160.114.04003 Boehringer Ingelheim Investigational Site, Zagreb
  - 1160.114.04004 Boehringer Ingelheim Investigational Site, Zagreb
- 1160.114.28001 Boehringer Ingelheim Investigational Site, Cairo, Egypt
- Germany (15):
  - 1160.114.490201 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.114.490216 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.114.490220 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.114.490217 Boehringer Ingelheim Investigational Site, Dessau
  - 1160.114.490214 Boehringer Ingelheim Investigational Site, Dinslaken
  - 1160.114.490215 Boehringer Ingelheim Investigational Site, Halle
  - 1160.114.490206 Boehringer Ingelheim Investigational Site, Itzehoe
  - 1160.114.490209 Boehringer Ingelheim Investigational Site, Kempen
  - 1160.114.490208 Boehringer Ingelheim Investigational Site, Ludwigsburg
  - 1160.114.490212 Boehringer Ingelheim Investigational Site, Markkleeberg
  - 1160.114.490207 Boehringer Ingelheim Investigational Site, Mühldorf
  - 1160.114.490210 Boehringer Ingelheim Investigational Site, München
  - 1160.114.490202 Boehringer Ingelheim Investigational Site, Northeim
  - 1160.114.490204 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1160.114.490211 Boehringer Ingelheim Investigational Site, Wittenberg
- 1160.114.07001 Boehringer Ingelheim Investigational Site, Beirut, Lebanon
- Netherlands (3):
  - 1160.114.31013 Boehringer Ingelheim Investigational Site, Deventer
  - 1160.114.31008 Boehringer Ingelheim Investigational Site, Enschede
  - 1160.114.31005 Boehringer Ingelheim Investigational Site, Maastricht
- Spain (9):
  - 1160.114.34012 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.114.34004 Boehringer Ingelheim Investigational Site, Jaén
  - 1160.114.34010 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.114.34003 Boehringer Ingelheim Investigational Site, Málaga
  - 1160.114.34005 Boehringer Ingelheim Investigational Site, Murcia
  - 1160.114.34013 Boehringer Ingelheim Investigational Site, Sabadell (Barcelona)
  - 1160.114.34011 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 1160.114.34001 Boehringer Ingelheim Investigational Site, Seville
  - 1160.114.34006 Boehringer Ingelheim Investigational Site, Seville
- Turkey (Türkiye) (4):
  - 1160.114.09004 Boehringer Ingelheim Investigational Site, Adana
  - 1160.114.09001 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.114.09006 Boehringer Ingelheim Investigational Site, Antalya
  - 1160.114.09009 Boehringer Ingelheim Investigational Site, Istanbul

REFERENCES:
- [Derived] Huisman MV, Lip GY, Diener HC, Dubner SJ, Halperin JL, Ma CS, Rothman KJ, Teutsch C, Zint K, Ackermann D, Clemens A, Bartels DB. Design and rationale of Global Registry on Long-Term Oral Antithrombotic Treatment in Patients with Atrial Fibrillation: a global registry program on long-term oral antithrombotic treatment in patients with atrial fibrillation. Am Heart J. 2014 Mar;167(3):329-34. doi: 10.1016/j.ahj.2013.12.006. Epub 2013 Dec 19. PMID 24576516

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 1063
Completed | 1063
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 1063
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486
  Male | 577

OUTCOME MEASURES:

1. Primary Outcome: CHADS2 Score
Description: CHADS2 score is based on a point system in which 2 points are assigned for a history of stroke or transient ischemic attack and 1 point each is assigned for age equal to or greater more than 75 years, hypertension, diabetes, or clinical heart failure or impaired left ventricular systolic function (generally interpreted as an ejection fraction ≤ 40%).
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  Low (Score=0) | 102
  Moderate (Score=1) | 386
  High (Score >=2) | 575

2. Primary Outcome: CHA2DS2-VASc Score
Description: The CHA2DS2-VASc risk score is based on a point system in which 2 points are assigned for a history of stroke or TIA, or age ≥75; and 1 point each is assigned for age 65-74 years, a hypertension, diabetes, cardiac failure, vascular disease and female sex. On the basis of the risk strata defined in previous guidelines, a CHA2DS2-VASc score of 0 corresponds to "low risk", a score of 1 corresponds to "intermediate risk", and a score of 2 or more corresponds to "high risk".
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  Low (Score=0) | 0
  Moderate (Score=1) | 226
  High (Score >=2) | 837

3. Primary Outcome: HAS-BLED Risk Score
Description: The HAS-BLED score is based on a point system in which 1 point is assigned for hypertension (systolic blood pressure >160 mmHg), 1 point for each of abnormal renal (presence of chronic dialysis or renal transplantation or serum creatinine ≥200 μmol/L) and liver (chronic hepatic disease or biochemical evidence of significant hepatic derangement) function, 1 point each is assigned for stroke, bleeding (previous bleeding history and/or predisposition to bleeding), labile Internation Normalized Ratios (INRs,unstable/high INRs or poor time in therapeutic range), age >65 years and 1 point each for drugs (such as antiplatelet agents, non-steroidal anti-inflammatory drugs) or alcohol.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  Low (Score <3) | 860
  High (Score >=3) | 121
  Missing | 82

4. Primary Outcome: Antithrombotic Treatment Choice at Baseline
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  None | 215
  Vitamin K Antagonist (VKA) | 349
  Acetylsalicylic Acid (ASA) | 443
  Antiplatelet agents other than ASA | 36
  Other | 20

5. Primary Outcome: Gender
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  Female | 486
  Male | 577

6. Primary Outcome: Age Group
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  <65 years | 382
  65 to <75 years | 314
  >= 75 years | 367

7. Primary Outcome: Medical History
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  Previous stroke | 110
  Coronary artery disease (CAD) | 256
  Congestive heart failure | 256
  History of hypertension | 795
  Diabetes mellitus | 240

8. Primary Outcome: Concomitant Medication
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1063
participants
  Antihypertensive/heart failure and antiarrhythmic | 739
  Metabolic and anti-inflammatory therapy | 395

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/1063
Other Adverse Events (participants affected / at risk) | 0/1063

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.